CLINICAL TRIAL: NCT05623202
Title: Pilot Intervention Study for Capacity-oriented Approaches to Food Security, Diet Quality, and Cardiovascular Disease Risk Among Hispanics/Latinos
Brief Title: Pilot Study of Capacity-oriented Intervention to Promote Food Security and Diet Quality Among Hispanics/Latinos
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HL150406
Record Dates: First submitted 2022-11-01; First posted 2022-11-21 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Nutrition, Healthy; Knowledge, Attitudes, Practice; Self Efficacy
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Capacity-oriented behavior-change intervention (Experimental)
  Interventions: Behavioral: Multi-level behavior-change intervention to strengthen food- and diet-related capital to promote food security and diet quality among low-income Hispanic/Latino adults

INTERVENTIONS:
Behavioral: Multi-level behavior-change intervention to strengthen food- and diet-related capital to promote food security and diet quality among low-income Hispanic/Latino adults — The behavior-change intervention with low-income Hispanic/Latino adults will mobilize existing sources of human, material, social, and cultural capital at the individual, household, social, and community level, and will include a nutrition education component and a food access component.

SUMMARY:
Despite a large proportion exhibiting cardiovascular disease risk factors and experiencing food insecurity, U.S. Hispanics/Latinos demonstrate low cardiovascular mortality, which may indicate existing capital (e.g., assets) protecting health and diet. The goal of this study is to evaluate the feasibility and short-term efficacy of a pilot intervention aimed at improving diet quality through strengthening food- and diet-related capital and food security among low-income, Hispanic/Latino adults in San Diego, California. The pilot intervention will be integrated into an existing local health or nutrition program serving low-income Hispanic/Latino adults. Participants will be asked to:

* Complete questionnaires before and after the intervention
* Engage in nutrition education activities
* Engage in food access-related activities

ELIGIBILITY:
Inclusion Criteria:

* Self-identified Hispanic/Latino
* Living full-time in San Diego County with no plan to move in next 3 months
* At or below 200% of Federal Poverty Line

Exclusion Criteria:

* Not Hispanic/Latino
* Living outside San Diego County
* Living only part-time in San Diego County
* Planning to move out of San Diego County in next 3 months
* >200% of Federal Poverty Line

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Diet quality | 3 months
  Food Behavior Checklist for Spanish-speaking participants

SECONDARY OUTCOMES:
Household food security status | 6 weeks, 3 months
  U.S. Department of Agriculture 18-item Household Food Security Survey Module
Self-efficacy for food security | 6 weeks, 3 months
  Self-efficacy for food security scale (Martin et al, 2016)
Food resource management knowledge | 6 weeks, 3 months
  Expanded Food and Nutrition Education Program (EFNEP) food resource management questionnaire
Food resource management knowledge | 6 weeks, 3 months
  Knowledge of available local food resources (checklist)
Food resource management skills | 6 weeks, 3 months
  Expanded Food and Nutrition Education Program (EFNEP) food resource management questionnaire
Food resource management skills | 6 weeks, 3 months
  Use/access of available local food resources (checklist)
Material capital | 6 weeks, 3 months
  Perceived neighborhood food availability and affordability scale
Human capital | 6 weeks, 3 months
  Life Orientation Test (optimism subscale)
Social capital | 6 weeks, 3 months
  Neighborhood cohesion scale
Social capital | 6 weeks, 3 months
  Family cohesion scale
Cultural capital | 6 weeks, 3 months
  Familism scale
Cultural capital | 6 weeks, 3 months
  Simpatia scale

IPD SHARING:
Plan to Share IPD: No